CLINICAL TRIAL: NCT00588458
Title: Primary Sclerosing Cholangitis: Value of Computerized Tomographic Cholangiography and Intraductal Volumetric Measurement in Determining the Prognosis
Brief Title: The Value of CT Cholangiography in Primary Sclerosing Cholangitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There is no participant enrolled in this study since developing this trial and other cholangiographic techniques are more available in our institute.
Sponsor: Mayo Clinic (Other)
Responsible Party: Phunchai Charatcharoenwitthaya, M.D., Mayo Clinic and Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06-002976 0
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary sclerosing cholangitis; Computed tomographic cholangiography; MELD score; Mayo risk score for PSC
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): All patients with PSC in will have CT cholangiography.
  Interventions: Procedure: CT cholangiography

INTERVENTIONS:
Procedure: CT cholangiography — Cholografin 20ml will be diluted in 100 ml of normal saline and infused over 30 minute time interval. Following the infusion of the cholografin, morphine (0.04 mg/kg) will be administered to contract the sphincter of Oddi and improve bile duct distension and visualization. Thirty minutes following the administration of morphine a test scan (CT cholangiography) will be performed through the liver to determine if there is adequate biliary excretion. The test scan will consist of 10 mm thick image obtained through the mid liver. If there is evidence of biliary excretion, high-resolution images will be performed through the liver and bile ducts. The axial images will be reconstructed into maximum intensity projection models and volume rendered models that can be viewed in 3-dimension.

SUMMARY:
The reason for this study is to see if a new radiologic technique called computerized tomographic cholangiography (CT cholangiography) could be helpful to demonstrate the bile ducts features and measure the amount of space of bile duct canals that should be filled with bile fluid. It may be useful to find out how well these findings correlate with the previously known clinical predictors in term of the clinical outcomes that will happen in the future for patients with primary sclerosing cholangitis (PSC).

DETAILED DESCRIPTION:
Prognostic models, which have been produced based on clinical, histological and biochemical feature, are useful in predicting survival and determining timing for liver transplantation. Preliminary feasibility studies in patients with PSC using high resolution CT with a contrast agent (CT cholangiography), has shown excellent depiction of bile ducts. CT cholangiography also has the potential to allow quantification of intraductal volume by using sophisticated computer programs. This assessment may be an important clinical feature to assess disease severity and progression.The information about cholangiographic features could be important for therapeutic decisions (e.g., in determining the usefulness of balloon dilatation or stenting for a dominant extrahepatic duct stricture), for counseling patients, and for therapeutic trials in stratifying patients and assessing efficacy of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females, age 18-70 (inclusive) with suspected PSC.
* Serum carbohydrate antigen 19-9 (CA19-9) level in normal range (obtained within the previous year), or if greater than normal, the patient requires a negative cytologic or histologic evidence for cholangiocarcinoma within prior 3 months.
* Sexually active female patients of childbearing potential must be evaluated for pregnancy. A pregnancy test obtained at entry prior to the initiation of treatment must by negative. Female patient must not be breast-feeding.
* Renal function: a creatinine less than 2.0 mg/dL or a diabetic patient with a creatinine less than 1.5 mg/dL.

Exclusion Criteria:

* Evidence of cholangiocarcinoma
* Pregnancy or breast feeding
* History of allergy to iodinated contrast agents or morphine
* Renal impairment as defined as known renal disease, a creatinine higher than 2.0 mg/dL or a diabetic patient with a creatinine higher than 1.5 mg/dL.
* Any known pre-existing medical condition that could interfere with the patient's participation in and completion of the study such as significant cardiovascular dysfunction or chronic obstructive pulmonary disease requiring specific therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
To determine the correlation between baseline characteristics of bile ducts and intraductal volume of the biliary tree by CT cholangiography and MELD score and the Mayo risk score in patients with PSC. | baseline

SECONDARY OUTCOMES:
To determine the correlation between change in characteristics of bile ducts and intraductal volume of the biliary tree by CT cholangiography and change in MELD score and the Mayo risk score after 2-years of follow-up as compared with baseline. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Phunchai Charatcharoenwitthaya, M.D., Principal Investigator — Mayo Clinic